CLINICAL TRIAL: NCT03375905
Title: Pilot Study to Evaluate the Effectiveness and Safety of the aerSleep™ System in an Ethnic Japanese Population Diagnosed With Obstructive Sleep Apnea (OSA)
Brief Title: Effectiveness and Safety of cNEP in Ethnic Japanese With Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sommetrics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOM-014
Record Dates: First submitted 2017-12-07; First posted 2017-12-18 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Obstructive Sleep Apnea
Keywords: ethnic Japanese
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- cNEP (Experimental): cNEP treatment
  Interventions: Device: cNEP

INTERVENTIONS:
Device: cNEP — subjects with OSA will be treated with the cNEP device with the goal of reducing the number of apneas and hypopneas
  Other Names: continuous negative external pressure

SUMMARY:
The aim of this study is to evaluate the effectiveness and safety of cNEP (continuous negative external pressure) for the treatment of obstructive sleep apnea during two weeks of home use in subjects of Japanese ethnicity.

ELIGIBILITY:
Inclusion Criteria:

* both parents ethnically Japanese, or one parent Japanese and the other east-Asian
* PSG (polysomnogram) done within the previous 12 months that shows an AHI of 10-50/hr and <80% of apneas and hypopneas are obstructive
* cNEP collar fits and is well-tolerated

Key exclusion Criteria:

* BMI >34
* abnormalities in neck structure
* sleep disturbance other than obstructive sleep apnea
* serious medical illness
* pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
proportion of sustained responders | two weeks after initiation of treatment
  reduction of AHI of >50% and to <15/hr from qualifying PSG

SECONDARY OUTCOMES:
proportion of initial responders | at PSG 1, one day
  reduction of AHI of >50% and to <15/hr from qualifying PSG
AHI comparison with qualifying PSG | one day, on three separate study occasions
  apnea-hypopnea index
ODI comparison with qualifying PSG | one day, on three separate study occasions
  oxygen desaturation index
SpO2 <90% comparison with qualifying PSG | one day, on three separate study occasions
  oxygen desaturation index <90%
CGI of sleep | three months, and two weeks, respectively
  clinical global impressions of sleep, comparing 3-month baseline with end of two weeks of treatment
CGI of satisfaction with the cNEP device | after two weeks of treatment
  clinical global impressions of the cNEP device
Treatment-emergent adverse events | two weeks
  tabulation of treatment-emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jamil S Sulieman, MD, Principal Investigator — The Sleep Lab, Kaneohe, HI
Locations (1):
- The Sleep Lab, Kaneohe, Hawaii, United States

IPD SHARING:
Plan to Share IPD: Undecided